CLINICAL TRIAL: NCT02816060
Title: Effectiveness of Neural Tensioner Exercise on Conditioned Pain Modulation, Disability and Range of Motion in Patients With Chronic Neck Pain: A Randomized Clinical Trial
Brief Title: Neural Tensioner Exercise on Conditioned Pain Modulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PT, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14/2013
Record Dates: First submitted 2016-06-09; First posted 2016-06-28 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Neck Pain; Diffuse Noxious Inhibitory Control
Keywords: pain measurement
MeSH Terms: conditions — Neck Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neural tensionner exercise (Experimental): This group will receive a specific tensionner nerve exercise to provide mechanical stress across the median nerve. This technique have two positions, start and end. It consists on going from one to the other position constantly, controlling the speed of the technique to be constant. In the start position, the subject will be supine lying on a couch with the following parameters: contralateral cervical side bending, shoulder depression, shoulder abduction and external rotation to 90°, elbow flexion to 90º, and forearm supination. In the final position, the therapist will perform full elbow extension while maintaining all the joints previously situated as described above until the patients feel tension, then return to the start position.
  Interventions: Procedure: manual therapy
- sham neural tensionner exercise (Placebo Comparator): The control group will receive a sham technique (ST) with minimal mechanical stress across the median nerve. Patients will be placed in neutral cervical spine position with no shoulder depression, shoulder abduction and external rotation to 45°, 45° of elbow extension, and forearm pronation.. This technique will be passively repeated from elbow flexion to extension in the same way than the NTE group
  Interventions: Procedure: manual therapy

INTERVENTIONS:
Procedure: manual therapy — manual therapy with neural exercise will be applied on patients with neck pain

SUMMARY:
Background: There is evidence linking conditioned pain modulation (CPM) deficiency with musculoskeletal pain syndromes such as fibromyalgia, migraine, tension-type headaches and irritable bowel syndrome, as well as with temporomandibular disorders, idiopathic facial pain and chronic fatigue syndrome. Evidence shows that in pre-surgical situations of chronic pain there is no activation of CPM.

Objectives: The purpose of this study is to measure the CPM response and determine whether neural tensioner exercise in patients with chronic neck pain is effective in the improvement of neck pain intensity, neck disability and cervical range of motion.

Design: Double-blind, randomized placebo clinical trial. Methods: Patients with neck pain will be randomly allocated into two groups: the neural tensionner exercise group (NTE) or the sham technique (ST) group.

Individuals will be included in the study if they meet the following inclusion criteria: aged 18-65 years, neck pain perceived in the posterior region of the cervical spine, from the superior nuchal line to the first thoracic spinous process with more than 12 weeks of evolution and without radicular symptoms radiated to the head. Neck pain intensity with a visual analogue scale (VAS), neck disability index (NDI), CPM, and cervical rang of motion will be measured pre and port intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-65 years.
* neck pain perceived in the posterior region of the cervical spine, from the superior nuchal line to the first thoracic spinous process with more than 12 weeks of evolution and without radicular symptoms radiated to the head, trunk, and/or the upper limbs.
* the ability to understand, write, and speak Spanish fluently

Exclusion Criteria:

* development of systemic or degenerative diseases;
* symptoms of depression according to Beck's questionnaire.
* pain in any area between the lower back and the head in the last 9 months.
* neck pain associated with whiplash injuries.
* medical red flag history (i.e., tumour, fracture, metabolic diseases, rheumatoid arthritis, osteoporosis). - neck pain with cervical radiculopathy.
* neck pain associated with externalized cervical disc herniation.
* fibromyalgia syndrome.
* previous neck surgery.
* neck pain accompanied by vertigo caused by vertebrobasilar insufficiency or accompanied by non-cervicogenic headaches due to a traumatic event in the past 12 months.
* and history of neck or face pain in the last 6 months.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Physiological parameter | 5 minutes
  Conditioned pain modulation: Diffusse noxious inhibitory control sistem will be measure with torniquete test

SECONDARY OUTCOMES:
Visual analogue scale | 5 minutes
  Neck pain intensity measured by visual analogue scale (VAS)
physiological movement | 5 minutes
  Cervical range of motion measured with cervical range of motion device

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández-Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez-Carnero J, Sierra-Silvestre E, Beltran-Alacreu H, Gil-Martinez A, La Touche R. Neural Tension Technique Improves Immediate Conditioned Pain Modulation in Patients with Chronic Neck Pain: A Randomized Clinical Trial. Pain Med. 2019 Jun 1;20(6):1227-1235. doi: 10.1093/pm/pny115. PMID 29945245
- See also: Related Info — http://www.urjc.es